CLINICAL TRIAL: NCT04510675
Title: A 6-Week, Randomized, Evaluator-Blinded, In Vivo Within Subject Repeat Test to Evaluate the Irritation and Sensitization Potential of Omeza Collagen Matrix in Healthy Volunteers
Brief Title: Irritation Potential of Omeza Collagen Matrix Using Modified HRIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omeza, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OMZRIP1F
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-02

CONDITIONS: Erythema; Sensitisation
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Intervention Model Description: The study design is based on a Modified Draize Human Repeat Insult Patch Test.
Masking Description: The trained skin evaluator and Investigator was blinded to the identity of the test materials. Test/control sites were randomized within participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test Article (Omeza Collagen Matrix) (Experimental): Repetitive and continuous patch applications of the test article to the same test sites on the back approximately 48 hours on weekdays and for approximately 72-hour periods over weekends over 3 weeks, for a total of 9 induction applications. During a subsequent challenge phase 10-17 days after the induction phase, the test article and negative control will be applied for 48 hours.
  Each subject will receive both the test article and negative control at the same time.
  Interventions: Device: Test Article
- Negative Control (0.9% aqueous sodium chloride) (Experimental): Repetitive and continuous patch applications of the negative control to the same test sites on the back approximately 48 hours on weekdays and for approximately 72-hour periods over weekends over 3 weeks, for a total of 9 induction applications. During a subsequent challenge phase 10-17 days after the induction phase, the test article and negative control will be applied for 48 hours.
  Each subject will receive both the test article and negative control at the same time.
  Interventions: Other: Negative Control

INTERVENTIONS:
Device: Test Article — Omeza Collagen Matrix
  Arms: Test Article (Omeza Collagen Matrix)
Other: Negative Control — Occlusive Patch of 0.9% sodium chloride, NaCl
  Arms: Negative Control (0.9% aqueous sodium chloride)

SUMMARY:
The primary objective of this study was to assess the sensitization potential of Omeza Collagen Matrix compared to that of a negative control based on a Modified Human Repeat Insult Patch Test.

ELIGIBILITY:
Inclusion Criteria:

* Good general health, as assessed by medical history and brief dermal skin examination of the application site (back);
* Was fully informed of the risks of entering the study and was willing to provide written consent to enter the study;
* Was willing to follow study rules, which included: no sun exposure (for example; no swimming, sunbathing, or tanning beds), avoided activities that would cause excessive sweating, abstained from use of lotions, creams, or oils on the back area;
* Was willing to not change current brand of personal care products such as soaps, body washes, laundry detergents, body sprays, body spritzes, etc. while participating on the study;
* Was willing and able to practice an acceptable measure of contraception (i.e. birth control medication for at least 3 months prior, condom with spermicide or birth control injections,) during the study, if female of childbearing potential. To be considered female of non-childbearing potential, subject must have had a hysterectomy, tubal ligation, or had been post-menopausal for at least 1 year.

Exclusion Criteria:

* Clinically significant skin disease which contraindicated participation, including psoriasis, eczema, atopic dermatitis, and active cancer;
* Asthma that required medication;
* Insulin-dependent diabetes;
* Known immunological disorders such as HIV positive, AIDS and systemic lupus
* erythematosus;
* Treatment for any type of cancer within the last six months;
* Routine use (as defined by using more than 3 days in a week) of any anti-inflammatory drug (e.g., aspirin, ibuprofen, corticosteroids; 81 mg aspirin is acceptable), immunosuppressive drugs, antihistamine medication (steroid nose drops and/or eye drops are acceptable) or over-the-counter pain medication that was ingested in quantities exceeding label instructions;
* Use of topical drugs at patch site;
* Pregnancy, lactation, or planning a pregnancy (confirmed by a urine pregnancy test administered to females of childbearing potential);
* Medical condition which, in the Investigator's judgement, made the subject
* ineligible or placed the subject at undue risk;
* Participation in any patch test for irritation or sensitization within the last four weeks;
* Dermatological aberrations in or around test sites which included sunburn, extremely deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or any other disfiguration of the test site;
* Confirmed allergy to adhesives, bandages, or ingredients in OmezaTM Collagen Matrix;
* History of anaphylaxis to matrix ingredients (e.g. fish, palm oil, hemp oil, beeswax).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Ellis, MD, Principal Investigator — PCR Corp; Lori DeCaro, Study Director — PCR Corp
Locations (1):
- PCR Corp, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Article (Omeza Collagen Matrix) and Negative Control (Occlusive Patch of 0.9% NaCl): Each subject will be treated with the test article (Omeza Collagen Matrix) and the negative control (Occlusive Patch of 0.9% sodium chloride, NaCl) at the same time.
  During an induction phase of the study, the test article and negative control will be applied repetitively and continuously on one side of the paraspinal region of the back. Each application will be for approximately 48 hours (weekdays) or 72 hours (weekends) over three weeks for a total of 9 applications. During a subsequent challenge phase 10-17 days after the induction phase, the test article and negative control will be applied for 48 hours. The application sites of subject will be evaluated using the Skin Irritation Scale at approximately 30 minutes, 24 hours, 48 hours, and 72 hours after removal of the test article and negative control.
Period: Overall Study
Arm/Group | Test Article (Omeza Collagen Matrix) and Negative Control (Occlusive Patch of 0.9% NaCl)
Started | 58
Completed | 53
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- Test Article and Control: Each subject will receive all investigational products at the same time.
  Test Article: Omeza Collagen Matrix
  Negative Control: Occlusive Patch of 0.9% sodium chloride, NaCl
Arm/Group | Test Article and Control
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 36
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Erythema During the Challenge Phase for Omeza Collagen Matrix
Description: Erythema is evaluated during the challenge phase based on a numeric scale from 0 - 3 (0: No visible reaction, +: Slight/patchy, 1: Mild, 2: Moderate, 3: Strong). A score of 1, 2, or 3 indicates dermal sensitization.
Time Frame: 24, 48, 72, and 96 Hours
Population: 58 subjects were enrolled with 53 subjects completing the study.
Measure: Count of Participants; unit: Participants
Groups:
- Test Article (Omeza Collagen Matrix): Repetitive and continuous patch applications of the test article (Omeza Collagen Matrix) to the same test sites on the back approximately 48 hours on weekdays and for approximately 72-hour periods over weekends over 3 weeks, for a total of 9 induction applications.
- Negative Control (0.9% Aqueous Sodium Chloride): Repetitive and continuous patch applications of the negative control (0.9% aqueous sodium chloride) to the same test sites on the back approximately 48 hours on weekdays and for approximately 72-hour periods over weekends over 3 weeks, for a total of 9 induction applications.
Arm/Group | Test Article (Omeza Collagen Matrix) | Negative Control (0.9% Aqueous Sodium Chloride)
Number analyzed (Participants) | 53 | 53
Participants
  Frequency of Irritation Score 0 at 24 Hours | 53 | 49
  Frequency of Irritation Score + at 24 Hours | 0 | 4
  Frequency of Irritation Score 1 at 24 Hours | 0 | 0
  Frequency of Irritation Score 2 at 24 Hours | 0 | 0
  Frequency of Irritation Score 3 at 24 Hours | 0 | 0
  Frequency of Irritation Score 0 at 48 Hours | 52 | 50
  Frequency of Irritation Score + at 48 Hours | 1 | 3
  Frequency of Irritation Score 1 at 48 Hours | 0 | 0
  Frequency of Irritation Score 2 at 48 Hours | 0 | 0
  Frequency of Irritation Score 3 at 48 Hours | 0 | 0
  Frequency of Irritation Score 0 at 72 Hours | 53 | 50
  Frequency of Irritation Score + at 72 Hours | 0 | 3
  Frequency of Irritation Score 1 at 72 Hours | 0 | 0
  Frequency of Irritation Score 2 at 72 Hours | 0 | 0
  Frequency of Irritation Score 3 at 72 Hours | 0 | 0
  Frequency of Irritation Score 0 at 96 Hours | 53 | 53
  Frequency of Irritation Score + at 96 Hours | 0 | 0
  Frequency of Irritation Score 1 at 96 Hours | 0 | 0
  Frequency of Irritation Score 2 at 96 Hours | 0 | 0
  Frequency of Irritation Score 3 at 96 Hours | 0 | 0

2. Secondary Outcome: Adverse Events Deemed Related to the Test Product or the Study
Description: The secondary outcome measure is the number of adverse events deemed related to the test article or the study.
Time Frame: 6 weeks
Population: While only 53 subjects completed the study, a total of 58 subjects were enrolled. Therefore, adverse events were assessed in relation to the entire 58 patients who were enrolled.
Measure: Number; unit: Adverse Events
Groups:
- Test Article (Omeza Collagen Matrix); Negative Control (Occlusive Patch of 0.9% NaCl): Each subject will be treated with the test article (Omeza Collagen Matrix) and the negative control (Occlusive Patch of 0.9% sodium chloride, NaCl) at the same time.
  During an induction phase of the study, the test article and negative control will be applied repetitively and continuously on one side of the paraspinal region of the back. Each application will be for approximately 48 hours (weekdays) or 72 hours (weekends) over three weeks for a total of 9 applications. During a subsequent challenge phase 10-17 days after the induction phase, the test article and negative control will be applied for 48 hours. The application sites of subject will be evaluated using the Skin Irritation Scale at approximately 30 minutes, 24 hours, 48 hours, and 72 hours after removal of the test article and negative control.
Arm/Group | Test Article (Omeza Collagen Matrix) | Negative Control (Occlusive Patch of 0.9% NaCl)
Number analyzed (Participants) | 58 | 58
Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study with each patient monitored over the 6 weeks of treatment.
Description: Since both the test article and negative control were administered at the same time, it would not be possible to determine if any systemic adverse events were related to the test article or the negative control. As such, the arms are combined for the adverse event record.
Groups:
- Test Article (Omeza Collagen Matrix) and Negative Control: Each subject was treated with the test article (Omeza Collagen Matrix) and the negative control (Occlusive Patch of 0.9% sodium chloride, NaCl) at the same time.
  During an induction phase of the study, the test article and negative control was applied repetitively and continuously on one side of the paraspinal region of the back. Each application was for approximately 48 hours (weekdays) or 72 hours (weekends) over three weeks for a total of 9 applications. During a subsequent challenge phase 10-17 days after the induction phase, the test article and negative control were applied for 48 hours. The application sites of subject were evaluated using the Skin Irritation Scale at approximately 30 minutes, 24 hours, 48 hours, and 72 hours after removal of the test article and negative control.
Arm/Group | Test Article (Omeza Collagen Matrix) and Negative Control
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 1/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Article (Omeza Collagen Matrix) and Negative Control (N=58)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Influenza deemed not related to the test article or negative control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT04510675/Prot_SAP_000.pdf